CLINICAL TRIAL: NCT01080495
Title: Evaluation of Radial Strain Versus Fractional Shortening and Fractional Area Change for Assessment of Left Ventricular Function in Transesophageal Echocardiography
Brief Title: Evaluation of Radial Strain for Assessment of Left Ventricular Function in Transesophageal Echocardiography
Acronym: Strain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Department of Anaesthesiology, Intensive Care and Pain Control, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 787/2009
Record Dates: First submitted 2010-02-11; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-02

CONDITIONS: Ventricular Function, Left
Keywords: left ventricular function; radial strain; fractional shortening; fractional area change
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEE (transesophageal echcardiography) (Other): all patients get TEE and all parameters (radial strain, fractional shortening and fractional area change) are evaluated
  Interventions: Procedure: TEE (transesophageal echocardiography)

INTERVENTIONS:
Procedure: TEE (transesophageal echocardiography) — a TEE is performed in all study objects and all parameters (radial strain, fractional shortening and fractional area change) are analysed
  Other Names: radial strain

SUMMARY:
Assessment of left ventricular function is an essential determinant of overall hemodynamics and heart function and therefore of central interest in intra-operative transesophageal echocardiography.

Currently, the most frequently used methods for quantification of left ventricular function are fractional shortening (FS) and fractional area change (FAC).

Radial strain is a new parameter to asses left ventricular function. The investigators want to assess left ventricular function with radial strain, fractional shortening (FS) and fractional area change (FAC) in non-cardiac patients during non-cardiac operations. The aim of this study is to show that radial strain is as reliable as FS and FAC in left ventricular function assessment and more robust to changes in preload and afterload conditions.

DETAILED DESCRIPTION:
Assessment of left ventricular function is an essential determinant of overall hemodynamics and heart function and therefore of central interest in intra-operative transesophageal echocardiography.

Currently, the most frequently used methods for quantification of left ventricular function are fractional shortening (FS) and fractional area change (FAC). These parameters can be assessed in the transgastric mid papillary short axis view (TG SAX) to quantify left ventricular systolic function. Limitations of these methods are the experience of the investigator - the more experienced the investigator the more reliable and reproducible the data are, load dependency of these methods and the geometrical assumption of a one-dimensional measurement for assessment of a three-dimensional contracting left ventricle. Therefore, LV-function will either be over- or underestimated by influence of segmental wall motion abnormalities or by missing them.

Radial strain allows reliable and reproducible evaluation of left ventricular function and also allows assessment of myocardial deformation from representative segments of each wall of the left ventricle. Myocardial strain is described as the relative deformation of a myocardial fiber, normalized to its original length:L1-L0/L0(%). Strain is positive (radial thickening) if L1>L0 and negative (longitudinal shortening and circumferential thinning) if L1<L0. Radial strain is sensitive to changes in contractility and less influenced by loading conditions which occur frequently during anaesthesia in a wide spectrum of non-cardiac surgery as a result of blood loss or loss of hemodynamic autoregulation due to anesthetic drugs.

Therefore we want to assess left ventricular function with radial strain, fractional shortening (FS) and fractional area change (FAC) in non-cardiac patients during non-cardiac operations. The aim of this study is to show that radial strain is as reliable as FS and FAC in left ventricular function assessment and more robust to changes in preload and afterload conditions.

Study hypothesis

The aim of the study is to compare fractional shortening (FS) and fractional area change (FAC) with radial strain from TG mid SAX using TEE in the anaesthetized patient undergoing non-cardiac surgery. Furthermore we want to investigate the influence of changes in loading conditions on these parameters in the anaesthetized non-cardiac patient undergoing non-cardiac surgery. Therefore patients are examined in zero position, trendelenburg- and anti-trendelenburg-position.

Hypothesis:

* Radial strain correlates with FAC and FS in assessment of left ventricular function in patients undergoing non-cardiac surgery. FAC is of primary interest because it has several advantages: it is very easy to calculate, it´s considered a surrogate of ejection fraction, and several studies have shown that it is an excellent measure of left ventricular function even in patients with heterogeneity of regional function.
* The parameters radial strain, fractional shortening and fractional area change correlate during are changes in loading conditions (zero-position, trendelenburg- and anti-trendelenburg-maneuver).

Study design: prospective cohort study Inclusion criteria

* Planned non-cardiac surgery with a minimum duration of 60 minutes, where intubation is indicated
* Age above 18 years
* Signed informed consent Exclusion criteria
* No patient's consent
* Subjects not able to understand study procedures
* Contraindications to transesophageal echocardiography (oesophageal-, gastric disorders, hematologic disorders with increased bleeding incidence, ENT-surgery, surgery of the oesophagus or stomach)
* Medical history of any kind of heart disease, dyspnea or angina pectoris
* Hypertension (medically treated)
* Diabetes
* Atrial fibrillation Study protocol One day prior to surgery the patients are screened and invited to participate in the study by the principle investigator. If they consent the principle investigator does a physical examination and takes their medical history.

On the day of surgery patients receive premedication as usual. Arriving at the operating room the patients are monitored with ECG, pulse oximetry and blood pressure (either invasive with insertion of an arterial catheter, when indicated, or non-invasive blood pressure). A peripheral venous line is needed for induction of anaesthesia. Induction and maintenance of anaesthesia is performed using standard protocols. After induction of anaesthesia and insertion of all needed catheters (central venous catheter, bladder catheter, arterial catheter, and eventually pulmonary artery catheter) the transoesophageal probe, covered with a special condom, will be inserted.

The examination will be done by the principle investigator (Dr. Ulrike Weber) under supervision of an expierenced investigator.

Intraoperative TEE-Examinations (T1, T2, T3)

At T1, T2, T3 TEE-study examinations are performed in zero position, Trendelenburg position, and anti-Trendelenburg position. Positioning will follow a random order according to a blinded randomization list.

Trendelenburg-position shall be defined for the study with 10cm head-down from horizontal position, anti-trendelenburg position with 10cm head-up (from horizontal position). After positioning examination will start after a 3 min delay for reaching a steady-state in loading conditions.

T1 - after induction of anesthesia

After insertion of the probe a transesophageal echo examination (TEE) is performed - including a complete routine clinical examination (T1):

T2 - Intraoperative TEE, 3min after positioning

Positioning (zero position, Trendelenburg, anti-trendelenburg) will be performed according to randomization. 3min after positioning, under stable hemodynamics, recordings of HR, blood pressure, FS, FAC, Radial strain

T3 - Intraoperative TEE, 3min after positioning

Positioning (zero position, Trendelenburg, anti-trendelenburg) will be performed according to randomization. 3min after positioning, under stable hemodynamics, recordings of HR, blood pressure, FS, FAC, Radial strain

The following measurements are taken for the study (3 times during sinus rhythm):

* FS in the transgastric short axis mid papillary view
* FAC in the transgastric short axis mid papillary view
* Radial strain in the transgastric short axis mid papillary view

Recordings of the 2D-mode images of the TG SAX shall be taken in triplicate with 3 heart cycles per stored clip. The images will be stored digitally in the EchoPAC-raw data format.

Analysis of data will be performed offline in a dedicated work station (EchoPAC, GE Vingmed, Horten, Norway). Three different investigators will analyse all data two times at two different time points.

Expected study population: 33 patients

ELIGIBILITY:
Inclusion Criteria:

* Planned non-cardiac surgery with a minimum duration of 60 minutes, where intubation is indicated
* Age above 18 years
* Signed informed consent

Exclusion Criteria:

* No patient's consent
* Subjects not able to understand study procedures
* Contraindications to transesophageal echocardiography (oesophageal-, gastric disorders, hematologic disorders with increased bleeding incidence, ENT-surgery, surgery of the oesophagus or stomach)
* Medical history of any kind of heart disease, dyspnea or angina pectoris
* Hypertension (medically treated)
* Diabetes
* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular function | 3min during TEE
  for left ventricular function transgastric short axis view is recorded 3 times for 3 heart cycles in 3 different positions (zero-position, trendelenburg- and antitrendelenburg-position)

SECONDARY OUTCOMES:
left ventricular function during changes in loading conditions | 3min during TEE
  for left ventricular function transgastric short axis view is recorded 3 times for 3 heart cycles in 3 different positions (zero-position, trendelenburg- and antitrendelenburg-position)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Department of Anaesthesiology, Intensive Care and Pain Control, University Hospital of Vienna
Locations (1):
- University Hospital of Vienna, Vienna, Vienna, Austria